CLINICAL TRIAL: NCT02302911
Title: Swiss Early Intervention Project in Autism: An Evaluation of Early Intervention Outcome
Acronym: SwissEIPA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: SWEIPA
Record Dates: First submitted 2014-10-23; First posted 2014-11-27 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Early intervention
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — no biospecimens are being retained
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Early intensive behavioral intervention: Children with a diagnosis of Autism Spectrum Disorder under the age of 5 years that are receiving early intensive behavioral Intervention at one of the participating centres.
  Interventions: Behavioral: Early intensive behavioral intervention
- Early intensive eclectic intervention: Children with a diagnosis of Autism Spectrum Disorder under the age of 5 years that are receiving early intensive eclectic Intervention at the participating centre.
  Interventions: Behavioral: Early intensive eclectic intervention
- Control group: Children with a diagnosis of Autism Spectrum Disorder under the age of 5 years that are receiving treatment as usual or no treatment at all.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Early intensive behavioral intervention — at least 10 hours a week of early intensive behavioral intervention
  Groups: Early intensive behavioral intervention
Behavioral: Early intensive eclectic intervention — at least 10 hours a week of early intensive eclectic intervention
  Groups: Early intensive eclectic intervention
Other: Treatment as usual — receipt of any Intervention that is less intensive than 10 hours a week
  Groups: Control group

SUMMARY:
This study aims to investigate the effectiveness of early (before the age of 5 years) and intensive intervention for children with Autism Spectrum Disorders.

DETAILED DESCRIPTION:
This study aims to investigate the effectiveness of early (before the age of 5 years) and intensive intervention for children with Autism Spectrum Disorders. The type of intervention proposed in Switzerland differs greatly depending on where people live. Several international studies show positive outcomes in children with Autism after receiving early behavioural intervention.

However, Disability Insurance (DI) in Switzerland does not fully cover these scientifically proven interventions. Since January 2014 they cover 45 000 CHF per child for only two years of early treatment across five centres chosen by the Federal Social Insurance Office. The remaining costs are covered by the parents, foundations or by the cantons. In addition, families benefit from this early intervention only if their child is enrolled in one of the five selected centres.

There are currently various types of support for children with Autism in Switzerland before age five, early intensive behavioural interventions, eclectic early intervention and less intensive interventions with a treatment that is not specific to Autism (about 3 hrs./week), which includes occupational therapy, speech therapy and early curative education. Some children do not receive any treatment.

This research aims to evaluate the efficacy of these interventions (early intensive behavioural/ eclectic/treatment as usual) as has been done previously in international studies. The study also aims to include centres other than those selected by the Swiss Federal Social Insurance Office.

ELIGIBILITY:
Inclusion criteria:

* For all groups:
* parents speak English, German or French
* diagnosis of Autism or Pervasive Developmental Disorder not otherwise specified
* 5 years or younger at the start of Intervention
* parents consent
* Experimental Group:
* family was accepted by one of the participating Service Providers

Exclusion Criteria:

* Experimental Group:
* receipt of a second intervention that either interferes with the intensive Intervention or is also intensive (more than 10 hours a week)
* Comparison Group:
* receipt of any Intervention that is more than 10 hours a week

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Experimental Groups: Child with Autism Spectrum Disorder diagnosis referred to one of the EIBI or EIEI Service Provider receiving Treatment as of January 2013.
  Control Group: Child with Autism Spectrum Disorder diagnosis receiving Treatment as usual and willing to participate
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2013-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Autism Diagnostic Observation Schedule-2 (ADOS-2) | Annually up to 3 years
  Measures autism symptom severity

SECONDARY OUTCOMES:
Positive Gain Scale | Annually up to 3 years
  Parent questionnaire
General Positive Affect Scale | Annually up to 3 years
  Parent questionnaire
Questionnaire on Resources and Stress | Annually up to 3 years
  Parent questionnaire
Hospital anxiety and Depression scale | Annually up to 3 years
  Parent questionnaire
Strengths and Difficulties Questionnaire | Annually up to 3 years
  Parent questionnaire to assess siblings' behavior and potential secondary effects of the intensive Intervention delivered
Vineland Adaptive Behavior Scales II (VABS) | Annually up to 3 years
  Parent interview; adaptive behavior
Snijders-Oomen nicht-verbaler Intelligenztest 2 1/2 - 7 (SON-R) | Annually up to 3 years
  IQ measure
Wechsler Preschool and Primary Scale of Intelligence-III (WPPSI-III) | Annually if child is testable up to 3 years
  IQ measure

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Gundelfinger, Dr. med., Principal Investigator — University of Zurich, Department of Child and Adolescent Psychiatry
Locations (3):
- Switzerland (3):
  - Autismuszentrum GSR, Aesch, Canton of Basel-City
  - Association Objectif Vaincre l'Autisme, Gland, Canton of Vaud
  - University of Zurich, Department of Child and Adolescent Psychiatry, Zurich